CLINICAL TRIAL: NCT05115773
Title: Comparison of The Effectiveness of Intraligamentary and Mandibular Anesthesia on Mandibular Molar Teeth: A Randomized Clinical Study
Brief Title: Comparison of The Effectiveness of Intraligamentary and Mandibular Anesthesia on Mandibular Molar Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Funda Cagırır Dindaroglu, Asst. Prof., Izmir Katip Celebi University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-TDU-DİŞF-0013
Record Dates: First submitted 2021-09-14; First posted 2021-11-10 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Anesthesia, Local
Keywords: intraligamentary anesthesia; inferior alveolar nerve block; paediatric dentistry

STUDY DESIGN:
Intervention Model Description: randomized controlled, single-blind, split-mouth clinical trial
Who Masked: Participant
Masking Description: Randomization was performed by a computer-generated random sorting sequence
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intraligamentary Anaesthesia (Experimental): Before the restorative treatment of mandibular first molar, SOPIRA® 30 gauge extra-short cartridge needle attached to the tip of the SOPIRA® Citoject (SOPIRA® Heraeus Kulzer, Hanau, Almanya) pressure injector will be inserted into the periodontal sulcus 1-2 mm until resistance. The needle will be at an angle of 30 degrees to the long axis of the tooth. As recommended by the manufacturer, a total of 0.36 ml (mesiobuccal and distobuccal) 4% articaine solution containing 1:100,000 epinephrine (Ultracaine DS forte cartridge, Sanofi-Aventis GmbH, Almanya) will be injected slowly over 42 seconds by pressing the dosing lever 3 times for each root. If the anaesthesia will be failed, we would use the 4-point IL injection by injecting the mesiolingual sulcus and distolingual sulcus with the same technique.
  Interventions: Procedure: Intraligamentary anaesthesia
- Mandibular Anaesthesia (Active Comparator): Before the restorative treatment of mandibular first molar, inferior alveolar nerve block will be provided using the direct standard method. The 27 gauge needle of a 2ml disposable plastic syringe (Ayset, Adana, Turkey) enters from the intersection of the internal oblique edge and the midline of the pterygomandibular raphe, and 1 ml of 4% articaine solution containing1:100,000 epinephrine (Ultracaine DS Forte ampul, Sanofi-Aventis GmbH, Almanya) will be injected slowly in 60 seconds. 15 minutes after the injection the anaesthesia of the lip/tongue will be checked by probing the labial mucosa of the ipsilateral canine tooth.
  Interventions: Procedure: Mandibular anaesthesia

INTERVENTIONS:
Procedure: Intraligamentary anaesthesia — one tooth anaesthesia by 2 or 4 points intraligamentary injection
  Other Names: 2 or 4 points intraligamentary injection
  Arms: Intraligamentary Anaesthesia
Procedure: Mandibular anaesthesia — Inferior alveolar nerve block by direct standart method
  Other Names: Inferior alveolar nerve block
  Arms: Mandibular Anaesthesia

SUMMARY:
This study aimed to compare the effects of mandibular and intraligamentary anesthesia techniques on pain scores during restorative treatment of permanent mandibular molars in pediatric patients. Additionally, comparing the anesthesia techniques in terms of injection pain, the success of anesthesia, postoperative complications, and the subjects' preference was planned.

This randomized, controlled, cross-over, single-blind, split-mouth study was conducted on 78 subjects aged 6 to 12 years. Subjects with enamel-dentin caries on the bilateral permanent mandibular molar were included.

DETAILED DESCRIPTION:
First, the subjects who met the inclusion criteria in the study were included in 2 study groups according to age, gender, dental experience, DMFT / dmft values, and ICDAS II and radiographic evaluation criteria. Two different anesthesia techniques were applied to the right / left permanent first molar teeth of the patients included in the study, with an interval of one week. The subjects have been divided into two groups as 39 subjects were Group 1 received intraligamentary anesthesia in the first visit, and 39 subjects were Group 2 received mandibular anesthesia in the first session. The pain perception rates of the patients during the injection and treatment phases were recorded subjectively using a visual analog scale and Wong-Baker FACES pain rating scale. Heart rate and arterial oxygen saturation were determined as the physiological parameters. The quality of anesthesia and success were evaluated by the operation at the end of each visit. Complications (pain, raised teeth, hematoma, trauma due to lip/tongue bites, swelling, infection, and bleeding) were explained to the patients after anesthesia. They were asked to take note of the complications they encountered. Postoperative complications were recorded by calling the cases 1 day after the 1st and 2nd visits. At the end of the second visit, anesthesia preference of the patient was asked and recorded.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with American Society of Anesthesiologists score I (ASA I)
* Subjects with Frankl's behavior rate III (positive) and IV (definitely positive),
* Subjects with indication of similar restoration treatment on bilateral first permanent mandibular molars
* Subjects whose plaque index score of 0 (no plaque) and 1
* Subjects whose gingival index score of 0

Exclusion Criteria:

* Allergic to the local anesthetics or sulfites
* Subjects with cholinesterase deficiency
* Subjects who use drugs that may affect the assessment of pain, such as narcotic or non-narcotic analgesic, anti-inflammatory, anxiolytic, antipsychotic and antihistamine agents
* Subjects who need to use sedatives or other medications during dental procedures

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 78 (Actual)
Dates: Start 2020-02-25 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
The measurements of dental pain using Visual Analogue Scale | Immediately after the working with a low-speed rotary instrument on dentin
  Subjective pain perception scores during the intervention using Visual Analogue Scale containing Numeric Rating Scale (0-10, where 0 means no pain/best, 10 - worst possible pain)
The measurements of injection pain using Visual Analogue Scale | Immediately after the local anaesthetic injection
  Subjective pain perception scores after the local anesthetic injection using Visual Analogue Scale containing Numeric Rating Scale (0-10, where 0 means no pain/best, 10 - worst possible pain)
Measurement of the pain perception during the dental procedures using Wong Baker FACES pain rating scale. | Immediately after the working with a low-speed rotary instrument on dentin
  Subjective pain perception scores using Wong Baker Faces pain rating scale (Face 0: it does not hurt/best, Face 2: it hurts a little, Face 4: it hurts a little more, Face 6: it hurts more, Face 8: it hurts a lot, Face 10: it hurts a lot/worst)
Measurement of the injection pain of the local anesthesia using Wong Baker FACES pain rating scale. | Immediately after the local anaesthetic injection
  Subjective pain perception scores using Wong Baker Faces pain rating scale (Face 0: it does not hurt/best, Face 2: it hurts a little, Face 4: it hurts a little more, Face 6: it hurts more, Face 8: it hurts a lot, Face 10: it hurts a lot/worst)
Change from baseline physiological parameters (arterial oxygen saturation and pulse rate) at the end of the working with a low-speed rotary instrument on dentin | Baseline and immediately after the working with a low-speed rotary instrument on dentin
  Measurement of arterial oxygen saturation and pulse rate using a pulse oximeter
Change from baseline physiological parameters (arterial oxygen saturation and pulse rate) at the end of the working with a low-speed rotary instrument on dentin | Baseline and immediately after the local anaesthetic injection
  Measurement of arterial oxygen saturation and pulse rate using a pulse oximeter
Practitioner's assessment of patient pain-related comfort | Immediately after the dental treatment
  Practitioner's subjective records: cases who need additional mandibular anaesthesia, whose treatment is completed without a discomfort related to pain, who has a slight discomfort even though additional mandibular anaesthesia is not needed during the treatment
Rate of post-op complication | Day after intervention
  Query the presence of post-op complications related to local anaesthesia

SECONDARY OUTCOMES:
Evaluate the correlation between two self reported objective pain scales | Immediately after the local anaesthetic injection
  The correlation between the scores of Wong Baker Faces pain rating scale (Face 0: it does not hurt/best, Face 2: it hurts a little, Face 4: it hurts a little more, Face 6: it hurts more, Face 8: it hurts a lot, Face 10: it hurts a lot/worst) and Visual Analogue Scale for pain (0-10, where 0 means no pain/best, 10 - worst possible pain) recorded after the local anaesthetic injection in 6-12 years old patients. For the Wong Baker FACES pain rating scale, the maximum value (10) means "it hurt a lot" is the worst and the minimum value (0) means "it does not hurt" is the best outcome. For the Visual Analogue Scale for pain containing Numeric Rating Scale , while the minimum value (0) means "no pain" is the best outcome, the maximum value (10) means "worst possible pain" is the worst outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Funda Çağırır Dindaroğlu, Asst. Prof., Study Director — İzmir Katip Çelebi University Faculty of Dentistry; Ece Yılmaz, DDS, Principal Investigator — Private Practice
Locations (1):
- Izmir Katip Celebi University, Izmir, Turkey (Türkiye)